CLINICAL TRIAL: NCT07226960
Title: Deprescribing in Outpatient Internal Medicine Practices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00137786
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Deprescribing
Keywords: Polypharmacy; medication regimens; medication reviews; geriatric patients
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Prospective, mixed methods, investigator-initiated pilot quality improvement analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medication review - deprescribing / de-escalation may occur (Experimental): Internal medicine providers and PharmDs will identify patients for whom a medication review and potential deprescribing / de-escalation intervention may be beneficial, and make recommendations to adjust therapy as appropriate.
  Interventions: Behavioral: medication review
- historical controls (No Intervention): No contact or intervention will be made with these patients, only retrospective chart review to gather data such as number of medications, hospitalizations, and falls. Patients included in the historical control arm will be matched to the intervention group based on sex, age, and number of medications as much as possible. The goal will be to include 50 patients in both the intervention and control arms.

INTERVENTIONS:
Behavioral: medication review — Internal medicine providers and PharmDs will identify patients for whom a medication review and potential deprescribing / de-escalation intervention may be beneficial.
  Other Names: potential deprescribing / de-escalation
  Arms: medication review - deprescribing / de-escalation may occur

SUMMARY:
The purpose of this study is to evaluate the impact of pharmacist-led medication reviews and deprescribing or de-escalation interventions on reducing the number of medications, falls, and hospitalizations, and improvement in quality of life in geriatric patients.

DETAILED DESCRIPTION:
With increasing age, key pharmacokinetic processes such as first-pass metabolism, bioavailability, drug distribution, and clearance, are affected, necessitating dose adjustments and careful medication management. Despite these risks, medication regimens in elderly patients are often left unchanged over time. Deprescribing, the intentional reduction or discontinuation of medications, has been shown to improve quality of life, reduce fall risk, minimize cognitive impairment, and decrease adverse drug interactions. In this analysis, the PharmD will perform a comprehensive medication review with the patient and collaborate with the provider and patient through shared decision making to deprescribe and/or dose reduce medication therapy where risks may outweigh benefits for the patient.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* taking 6 or more medications

Exclusion Criteria:

* patients in hospice or palliative care
* in Skilled Nursing Facility
* receiving cancer/oncology treatment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in number of medications | Month 3
  Change in number of medications

SECONDARY OUTCOMES:
Change in Medication Appropriateness Index scores | Month 3
  The Medication Appropriateness Index (MAI) score is a quantitative measure of prescribing appropriateness, where lower scores indicate more appropriate medication use, and higher scores indicate less appropriate use.
  Each criterion is rated on a 3-point scale:
  Appropriate (score of 0 or a low value) Each criterion is assigned a weight ranging from 1 to 3, with a maximum total score of 18 possible per drug.
  A summated score can be calculated for a patient by combining the scores for all their medications. This summated score is not standardized, meaning the potential total score depends on the number of medications the patient is taking. A score of 0 for a medication indicates ideal or appropriate prescribing for that specific criterion. Higher scores are associated with potentially inappropriate medication (PIM) use, increased risk of adverse drug events (ADEs), higher rates of unscheduled ambulatory or emergency department visits, and lower health-related quality of life.
Change in Quality of life scores | Month 3
  The Lübeck Medication Satisfaction Questionnaire (LMSQ) is scored by calculating the average score for each of its six subscales, which are based on three Likert-scale items each. Patients rate their agreement with each statement on a four-point scale (1=strongly disagree, 4=strongly agree), but items phrased negatively must be reverse-scored before calculating the subscale average. To get the subscale score, you sum the three items' scores and divide by three.
Number of documented falls | Month 3
  Number of documented falls
Number of documented hospitalizations | Month 3
  Number of documented hospitalizations
Number of documented visits to Primary Care Physician office | Month 3
  Number of documented visits to Primary Care Physician office

OTHER OUTCOMES:
Number of Pharmacist interventions | Month 3
  Documented via Medication therapy problems (MTP) tracking -

CONTACTS AND LOCATIONS:
Overall Officials: Julia Clements, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No